CLINICAL TRIAL: NCT05075525
Title: EFFECT OF HIGH INTENSITY LASER THERAPY ON PAIN AND LOWER EXTREMITY FUNCTION IN PATELLOFEMORAL PAIN SYNDROME
Brief Title: EFFECT OF HIGH INTENSITY LASER IN PATELLOFEMORAL PAIN SYNDROME
Acronym: Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ozluozge, Principal Investigator, MSc, PT, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ozgeozlu
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Physical Therapy; Orthopedic Disorder
Keywords: Patellofemoral pain; High intensity laser therapy
MeSH Terms: conditions — Musculoskeletal Diseases; Patellofemoral Pain Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to allocation and outcomes measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Laser Therapy Group (Experimental): Patients underwent High Intensity Laser Therapy (HILT) and exercise for 10 sessions
  Interventions: Other: High Intensity Laser Therapy Group
- Ultrasound and Transcutaneous Electrical Nerve Stimulation Group (Experimental): Patients will be treated by transcutaneous electrical nerve stimulation(TENS), ultrasound (US) and exercise for 10 sessions
  Interventions: Other: Ultrasound and Transcutaneous Electrical Nerve Stimulation Group
- Ultrasound and Interferential Current Stimulation Group (Experimental): Patients will be treated with ultrasound (US) ,interferential current stimulation and exercise for 10 sessions
  Interventions: Other: Ultrasound and Interferential Current Stimulation Group

INTERVENTIONS:
Other: High Intensity Laser Therapy Group — High Intensity Laser Therapy (HILT) and exercises will be used.
  Arms: High Intensity Laser Therapy Group
Other: Ultrasound and Transcutaneous Electrical Nerve Stimulation Group — Transcutaneous electrical nerve stimulation(TENS), ultrasound (US) will be applied.
  Arms: Ultrasound and Transcutaneous Electrical Nerve Stimulation Group
Other: Ultrasound and Interferential Current Stimulation Group — Ultrasound (US) ,interferential current stimulation and exercise will be used.
  Arms: Ultrasound and Interferential Current Stimulation Group

SUMMARY:
The aim of this study is to investigate the effectiveness of high-intensity laser therapy on pain and lower extremity function in the treatment of patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Participants between the ages of 25-45 who were diagnosed with Unilateral patellofemoral pain syndrome by the doctor will be included in the study. Also positive Clarke's test and patellar compression tests will be determined as inclusion criteria. The 45 participants will be randomly divided into three groups. Both groups will receive 2 weeks (5 sessions per week) of therapy. First group patients underwent High Intensity Laser Therapy (HILT) and exercises. Second group patients will be treated by transcutaneous electrical nerve stimulation(TENS), ultrasound (US) and exercise for 10 sessions. Also In the third group patients will be treated with ultrasound (US),interferential current stimulation and exercise. All groups receive the same exercise exercise protocol including muscle strengthening and flexibility training for 12 weeks. The outcomes will be pain intensity measured by visual analog scale (VAS) , knee flexion range of motion (FROM), timed up and go test (TUG),muscle strength measured with handheld dynamometer, Pressure Pain Threshold with an algometry and functionality of knee measured by the Lower extremity functional scale and Kujala patellofemoral questionnaire. Statistical analyzes will be performed to compare amounts at baseline, immediately after treatment, and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral patellofemoral pain syndrome diagnosed by a doctor
* 25-45 years old
* pain from prolonged sitting, climbing and descending stairs, running,knee bend more than 3 months
* positive patellar compression and clarke's tests.

Exclusion Criteria:

* Previous knee pain, trauma, surgery and other joint diseases,
* Knee ligament, bursa, meniscus and synovial fold injury or dysfunction
* Osteoarthritis in the knee joint,
* Neurological problems that may affect walking
* Pregnancy
* No chronic disease
* Malignancy,
* Presence of infection

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-03-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Pain status | 5 minutes
  Pain intensity was evaluated with visual analog scale (VAS) in two conditions during activity and resting time. This method, which is developed to determine the intensity of pain to indicate by numbers. It begins with the absence of pain (0) on numerical scale and ends the level of unbearable pain
Range of motion assesment | 10minutes
  Universal goniometer will used to measure the joint position and joint range of motion measurements based on Kendall and American Association of Orthopedic Surgeons. The participant will in the sitting position and asked to perform active cervical region flexion, extension, right and left rotation, right and left lateral flexion of the neck movements and performed degrees will recorded
Functionality | 5 minutes
  The patients will asked to start from a sitting position in a chair, to get up at the command given, to walk the predetermined distance of 3 meters as fast as they could, and to return to their seats. The time from the time they got up from the chair and sat down again will recorded with a stopwatch. Measurements will be repeated 3 times and the average will be recorded in seconds (sec).
Muscle stength assesment | 10 minutes
  A myometer will be used to measure the strength of the hamstring and quadriceps muscle groups of all participants. Myometer is an evaluation method that objectively evaluates muscle strength and gives more sensitive results than manual muscle testing.
Pain threshold assessment | 10 minutes
  Pressure pain threshold measurement will be measured with an algometer device. Algometers are a device that can be used to define pressure and pressure pain threshold.
Severity and function of patellofemoral pain | 5 minutes
  It will be evaluated with the 'Kujala patellofemoral score' system. These scoring system values range from 100 (normal, pain-free, fully functional knee) to 0 (severe knee pain and dysfunction).
Function of lower extremity | 10 minutes
  A lower extremity function test will be used to measure lower extremity functionality. It is a test used to measure the functional status of the lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: OZGE OZLU, Principal Investigator — Medipol University
Locations (1):
- Ozge Ozlu, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When I published this manuscript in a journal, I would share the results of inividuald participant data of this study with other researchers.

REFERENCES:
- [Result] Nazari A, Moezy A, Nejati P, Mazaherinezhad A. Efficacy of high-intensity laser therapy in comparison with conventional physiotherapy and exercise therapy on pain and function of patients with knee osteoarthritis: a randomized controlled trial with 12-week follow up. Lasers Med Sci. 2019 Apr;34(3):505-516. doi: 10.1007/s10103-018-2624-4. Epub 2018 Sep 3. PMID 30178432